CLINICAL TRIAL: NCT07168889
Title: The Choice of Mitral Valve Surgery Type and Mid-term Outcomes in Patients up to 70-years: Results of the AUTHEARTVISIT Study
Status: Completed | Type: Observational
Sponsor: Alissa Florian (Other)
Responsible Party: Sponsor-Investigator, Alissa Florian, Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: GS1-EK-4/722-2021-2
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mitral Valve Replacement
Keywords: mitral valve; bioprostheses; mechanical prostheses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBMVR: biological mitral valve replacement
- SMMVR: mechanical mitral valve replacement

SUMMARY:
The goal of this observational study is to learn about the long-term effects of mechanical versus biological mitral valve replacement in patients aged 70 years or younger. The main question it aims to answer is:

Do patients who receive a mechanical mitral valve live longer and need fewer repeat operations compared with those who receive a biological valve? Participants are patients in Austria who already had mitral valve surgery between 2010 and 2020 as part of their regular medical care. Information about their surgeries, health conditions, and outcomes was collected from national health insurance records. Researchers will follow these patients for up to 10 years to compare survival, reoperation rates, and other heart-related events between mechanical and biological valve recipients.

DETAILED DESCRIPTION:
This nationwide, registry-based, retrospective cohort study is part of the AUTHEART VISIT project, which investigates long-term outcomes of cardiac surgery in Austria. The present analysis focuses on patients aged 70 years or younger undergoing surgical mitral valve replacement (MVR) between January 1, 2010 and December 31, 2020. The aim is to evaluate differences in survival, reoperation rates, and cardiovascular outcomes between patients receiving mechanical mitral valve replacement (SMMVR) and those receiving biological mitral valve replacement (SBMVR).

Data source and registry procedures:

Data were obtained from the Austrian Health Insurance Funds, which cover approximately 98% of the Austrian population. The registry includes detailed patient-level information on diagnoses, procedures, and outcomes based on mandatory coding for reimbursement (ICD-10 for diagnoses and MEL codes for surgical procedures). The data are anonymized prior to analysis.

Quality assurance:

Data integrity is ensured by several mechanisms:

Data validation: Automatic data checks are performed to confirm plausibility, completeness, and consistency with predefined coding rules.

Source verification: Information is cross-checked against external records where available (e.g., insurance billing and hospital discharge data).

Data dictionary: A standardized coding framework is maintained, including MEL codes for procedures and ICD-10 for diagnoses. Definitions of outcomes are harmonized with prior AUTHEART VISIT studies.

Standard operating procedures: Established registry protocols govern data management, statistical analysis, and reporting.

Sample size and follow-up:

The study population includes all eligible patients undergoing mitral valve surgery in Austria during the study period (N=3520), with 413 undergoing sM-MVR, 487 undergoing sB-MVR, and 2620 undergoing mitral valve repair (MVRe). Median follow-up times were 6.6 years for SMMVR, 7.4 years for SBMVR, and 5.8 years for MVRe.

Handling of missing data:

Cases with implausible entries (e.g., death date before index surgery) are excluded. Missing values in baseline covariates are addressed through exclusion or handled in the propensity score weighting model. Outcome variables are based on administrative coding, minimizing missingness.

Statistical analysis plan:

The primary outcome is all-cause mortality. Secondary outcomes include reoperation, reoperation-free survival, major adverse cardiac events (MACE), myocardial infarction, heart failure, stroke, and bleeding. Time-to-event analyses are conducted using Cox proportional hazards models adjusted for age, sex, comorbidities, and concomitant procedures. To account for potential imbalances between groups, inverse probability of treatment weighting (IPTW) is applied based on a multinomial logistic regression model. Weighted and unweighted Kaplan-Meier curves are generated, with subgroup analyses by age. Cause-specific hazard models are used for secondary outcomes. Proportional hazards assumptions are evaluated using Schoenfeld residuals. A p-value <0.05 is considered statistically significant.

This registry-based approach provides comprehensive, real-world evidence on prosthesis choice in surgical MVR, with rigorous quality assurance procedures to ensure reliability and generalizability of results.

ELIGIBILITY:
Inclusion Criteria:

* Mitral valve surgery between 01.01.2010 and 31.12.2020

Exclusion Criteria:

* concomitant procedures on other valves

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Austria. The data included 3,520 patients aged ≤70 years who underwent mitral heart valve surgery between 1.1.2010 and 31.12.2020 in Austria.
Sampling Method: Non-Probability Sample
Enrollment: 3520 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
all-cause death | 10 years
  rate of all-cause death

SECONDARY OUTCOMES:
major adverse cardiac events | 10 years
  rate of major adverse cardiac events
reoperation-free survival | 10 years
  rate of reoperation-free survival
reoperation | 10 years
  rate of reoperation
myocardial infarction | 10 years
  rate of myocardial infarction
heart failure | 10 years
  rate of heart failure
stroke | 10 years
  rate of stroke
intracerebral hemorrhage | 10 years
  rate of intracerebral hemorrhage
bleeding other than ICH | 10 years
  rate of bleeding other than ICH

IPD SHARING:
Plan to Share IPD: No